CLINICAL TRIAL: NCT04590274
Title: Safety and Efficacy of Hydroxychloroquine for the Treatment & Prevention of Coronavirus Disease 2019 (COVID-19) Caused by Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Investigative Team no longer interested
Sponsor: International Brain Research Foundation (Other)
Responsible Party: Principal Investigator, Philip DeFina, PhD, Chief Executive Officer, International Brain Research Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CTP-HCQ-COVID19
Record Dates: First submitted 2020-10-07; First posted 2020-10-19 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Covid19; SARS (Severe Acute Respiratory Syndrome)
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome | interventions — Hydroxychloroquine; Vitamins; Minerals; Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Regimen (Experimental): 0-400 mg Hydroxychloroquine 0-500 mg Azithromycin 0-50 mg elemental Zinc 0-3,000 mg Vitamin C 0-5,000 IU Vitamin D3 0-1200 mg N-acetylcysteine 0-600 mg Elderberry 0-600 mg Quercetin
  Interventions: Drug: Hydroxychloroquine; Dietary Supplement: Vitamins and Minerals; Drug: Azithromycin

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine
Dietary Supplement: Vitamins and Minerals — elemental Zinc Vitamin C Vitamin D3 N-acetylcysteine Elderberry Quercetin
Drug: Azithromycin — Azithromycin

SUMMARY:
Coronavirus Disease 2019 (COVID-19) (previously called 2019-nCOV acute respiratory disease) is caused by SARS-CoV-2, a positive-sense single-stranded RNA virus of the coronavirus family. The coronaviruses are largely responsible for the common cold, the 2002 SARS outbreak in Guangdong, China, the 2012 MERS outbreak in Saudi Arabia, and the present COVID-19 outbreak that originated in Wuhan, China. Much has been reported by way of systemic injury caused by COVID-19 affecting the cardiovascular, hepatic, nervous systems. These conditions are likely the result of the virus overwhelming the immune system. For these reasons, the investigators wish to conduct this study using existing medications off-label, and over-the-counter supplements to support the immune response, prevent lasting injury, and hasten the recovery from COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1) Patients must have one or more of the following:

1. confirmed diagnosis of active SARS-CoV-2 infection, diagnosed with PCR
2. continued close contact with an individual with suspected SARS-CoV-2 infection
3. at risk for SARS-CoV-2 infection in the opinion of the treating physician or Principal Investigator.

Exclusion Criteria:

1) Patients must not have any uncontrolled disease such as:

1. cardiovascular disease
2. hepatic disease
3. renal disease
4. metabolic disease
5. other diseases or insufficiencies

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of individuals who develop COVID-19 symptoms | 6 months from study start
  The investigators will compare what percentage of participants in this study go on to develop COVID-19 symptoms, as compared to individuals not on the medicational regimen in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Philip DeFina, PhD, Principal Investigator — International Brain Research Foundation